CLINICAL TRIAL: NCT03971929
Title: A Phase I, Randomized, Double-Blind, Placebo-hydrochlorothiazide Parallel Controlled, Multiple-Ascending Dose Study to Evaluate the Safety, Efficacy of SHR 0532 Oral Tablets in Mild Hypertension Subjects
Brief Title: Safety and Effect Study of SHR0532 (Drug Code) Tablets in Patients With Mild Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR0532-102
Record Dates: First submitted 2019-05-28; First posted 2019-06-03 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2019-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR0532 tablet (Experimental): up to 3 cohorts of subjects will receive multiple dose of oral tablets
  Interventions: Drug: SHR0532
- SHR0532 placebo (Placebo Comparator): up to 3 cohorts of subjects will receive multiple dose of oral SHR0532 placebo
  Interventions: Drug: SHR placebo
- Hydrochlorothiazide (Active Comparator): up to 3 cohorts of subjects will receive multiple dose of oral Hydrochlorothiazide 25mg
  Interventions: Drug: Hydrochlorothiazide 25 mg

INTERVENTIONS:
Drug: SHR0532 — once daily(QD) for 4weeks
  Arms: SHR0532 tablet
Drug: SHR placebo — once daily(QD) for 4weeks
  Arms: SHR0532 placebo
Drug: Hydrochlorothiazide 25 mg — once daily(QD) for 4weeks
  Arms: Hydrochlorothiazide

SUMMARY:
The study is being conducted to evaluate the safety and efficacy and Pharmacokinetics/Pharmacodynamics of SHR0532 in subjects with mild hypertension for 4 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multiple ascending dose, placebo- and Hydrochlorothiazide-controlled study to evaluate the safety and tolerability, Pharmacokinetics and Pharmacodynamics and effect on blood pressure of SHR0532 tablets in patients with mild hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 to 65 years old
* Diagnosis of mild hypertension
* 18.5 kg/m2≤Body mass index (BMI) ≤35 kg/m^2
* Understand the study procedure and method, willing to participate the study and Informed consent form (ICF) signed in writing

Exclusion Criteria:

* History of significant drug allergy or allergic diseases (asthma, urticaria, eczematous dermatitis), or known allergy to anti hypertension drugs
* Anti-hypertensive drugs were taken within 1 month before screening
* History or at present patient has orthostatic hypotension
* History or at screening Participant has plasma sodium lower than 135mmol/L
* History or at screening visit/baseline patient has elevated serum uric acid (serum uric acid higher than ULN)
* Patients with type 1 diabetes mellitus need insulin therapy or poor blood glucose control (HbA1c > 9%, or oral anti diabetic drug dosage is not stable within 4 weeks before screening)
* History of arrhythmia or patient has clinically significant abnormalities of 12-lead ECG or prolonged corrected QT (QTc) interval (male > 450ms; female > 460ms) at screening visit
* History of New York Heart Association (NYHA) Definition II-IV Heart Failure
* Severe cardiovascular diseases occurred within 6 months before screening, including ischemic heart disease, peripheral vascular disease, significant ventricular tachycardia, atrial fibrillation, atrial flutter or other serious arrhythmias, hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, aortic or mitral valve disease of great hemodynamic significance, and severe cerebrovascular disease
* History of percutaneous intervention (PCI) or coronary artery bypass graft (CABG)
* History or active stroke, chronic seizures, or major neurological disorder
* History of osteoporosis, nephrocalcinosis, nephrolithiasis or hypercalciuria
* History or active malignant neoplastic disease. Exceptions: malignancies which have been successfully treated and non-recurrence >10 years prior to the screening visit
* Patients having following diseases may affect drug absorption, distribution, metabolism and excretion:

Gastrointestinal diseases such as irritable bowel syndrome, inflammatory bowel diseases including ulcerative colitis, Crohn's disease, malabsorption syndrome, microbial dysbiosis, intestinal infection; History of gastrointestinal operations, such as gastric resection and bypass, small intestinal resection and colonic resection which may affect drug absorption

* History of acute or chronic kidney diseases
* Dehydration or volume-depletion
* Clinically significant chronic or acute infectious diseases occur within 2 weeks before the start of the study (enrolment);
* Major surgery within 3 months before dosing
* Donation of blood/plasma within 1 month before dosing or blood/plasma (≥400 mL) within 3 months before dosing
* Unstable or severe urinary, digestive, psychiatric, neural, hematological and other diseases, or lab abnormalities, the investigators determine that participants in the study will be at unacceptable risk

Taking or having the following medication history:

* Participant need taking Cytochrome P450 3A4 (CYP3A4) inhibitors (such as ritonavir, indinavir, nelfinavir, erythromycin, telithromycin, clarithromycin, chloramphenicol, fluconazole, ketoconazole, itraconazole, verapamil or diltiazem) as well as strong/moderate CYP3A4 inducers (such as phenytoin, carbamazepine, oxcarbazepine, phenobarbital, efavirenz, nevirapine, rifampicin, modafinil, cyproterone or progestin) at least 2 weeks or 5 half-lives prior to administration of the initial dose of study drug until the post study visit
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) at least 2 weeks before 1st dose of study drug until the post study visit
* use of systemic glucocorticoid therapy

Any laboratory examination result meet the following criteria at screening/baseline:

* Serum potassium < 3.5mmol/L or > 5.5mmol/L
* Serum creatinine more than ULN, Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) more than 2.0 x ULN or total bilirubin more than 1.5 x ULN at screening/baseline visit
* Creatinine kinase (CK) more than 3.0 x ULN at screening/baseline visit;
* Clinically significant abnormalities of coagulation and thyroid function
* HbsAg and Hepatitis B Virus (HBV)-DNA> 1000 cps/ml, Hepatitis C Virus Antibody (HCVAb), syphilis and HIV antibodies were positive at screening visit
* Serum pregnant test positive at screening/baseline visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Adverse Events(AEs) and Serious Adverse Events （SAEs） | from informed consent form signature to the end of the study (up to 2 months)
  Incidence of AEs and SAEs, incidence of Treatment-Emergent Adverse Events, incidence of drug related adverse events (safety and tolrability)

SECONDARY OUTCOMES:
Change From Baseline in Clinic Systolic Blood Pressure (SBP) and Clinic Diastolic Blood Pressure (DBP) | Baseline to end of the study (up to 32 days)
  Each subject has their office blood pressure every day of each treatment period (total of 28 days of treatment). The difference between baseline and D28 of each office BP value are calculated and recorded.
Change from baseline in 24h Urine sodium | from baseline to Day 8; from D28 to D32 (up to 32 days)
  Urine sodium (Na) levels were measured over 24-hours and different time period of 24 hours on Day -1 (baseline) and on Day 1to Day 7, Day28 to Day 32. The total amount of Na excreted in the Urine for Day-1 (baseline) and Day1 to Day 7, Day 28 to Day 32 were calculated and recorded and the difference between the 2 values are recorded.
Change from baseline in 24h Urine Volume | from baseline to Day 8; from D28 to D32 (up to 32 days)
  Urine Volume were measured over 24-hours and different time period of 24 hours on Day -1 (baseline) and on Day 1to Day 7, Day28 to Day 32.The total amount of Urine excreted for Day-1 (baseline) and Day1 to Day 7, Day 28 to Day 32 were calculated and recorded and the difference between the 2 values are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided